CLINICAL TRIAL: NCT04918368
Title: Do Low Vitramin D Levels Increase the Frequency of Sleep Disorders and Anxiety in the 2nd and 3rd Trimester?
Brief Title: Vitamin D and Sleep Disorders in Pregnancy
Status: Completed | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Fatma ketenci gencer, Dr., Gaziosmanpasa Research and Education Hospital
Other Study IDs: GaziosmanpasaTREHc
Record Dates: First submitted 2021-04-17; First posted 2021-06-08 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2018-04

CONDITIONS: Sleep Disorder; Pregnancy Related; Vitamin D Deficiency
Keywords: anxiety; Pregnancy,; Sleep Wake Disorders; Vitamin D
MeSH Terms: conditions — Sleep Wake Disorders; Vitamin D Deficiency; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women between 18-45 years old, being in second and third trimester of a singleton pregnancy
  Interventions: Behavioral: Behavioral scales were used

INTERVENTIONS:
Behavioral: Behavioral scales were used — Women's Health Initiative Sleeplessness Scale (WHISS) and State Anxiety Scale (SAS), were applied.

SUMMARY:
Lack of sleep and poor sleep quality in pregnant women are associated with maternal depression and cognitive-sensual irregularities. These irregularities were reported worsening women's life quality and even increasing suicide ideation. It is also associated with obstetrical complications such as fetal growth deficiency, preterm birth, prolonged labor, preeclampsia and increased abdominal delivery frequency.Vitamin D also may affect the sleep indirectly through the cases with nonspecific pains. It was reported that vitamin D levels are correlated with sleep disorders such as obstructive sleep apnea and restless legs syndrome. The primary purpose of this study is to examine sleep disorders and vitamin D levels in pregnant women, and also, secondarily, vitamin D - anxiety and sleep disorders - anxiety relations were assessed.

ELIGIBILITY:
Inclusion Criteria:

* singletone pregnant women
* second and third trimester pregnant women

Exclusion Criteria:

* psychiatric disorder
* sleep disorder

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 225 pregnant women who are in second or third trimester of pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2017-08-20 (Actual); Primary Completion 2018-12-25 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Health Initiative Sleeplessness Scale (WHISS) | Through study completion, an average of 1 year
  Women's Health Initiative Sleeplessness Scale (WHISS) was used to assess the sleep status of pregnant women. In this scale consisting of five questions, first four questions focus on the period of time when sleeplessness started, status of not being able to continue the sleep and waking up early in the morning, while the last one focusses to determine the sleep quality. Scores of the scale range between 0 - 20. A score equal and above 10 means a sleeplessness problem. An increase in score means intensifying the sleeplessness symptoms.
State Anxiety Scale (SAS) | Through study completion, an average of 1 year
  In anxiety screening of pregnant women, State Anxiety Scale (SAS) was used. Scores of the scale including twenty questions range between min. 20 and max. 80. Higher scores mean higher anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Fatma Ketenci Gencer, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No